CLINICAL TRIAL: NCT01796249
Title: Prediction of Immediate Postoperative Pain Using Analgesia/Nociception Index (ANI): an Observational Study
Brief Title: Prediction of Immediate Postoperative Pain Using Analgesia/Nociception Index (ANI)
Status: Completed | Type: Observational
Sponsor: Emmanuel Boselli (Other)
Responsible Party: Sponsor-Investigator, Emmanuel Boselli, MD, PhD, Hôpital Edouard Herriot
Organization: Hôpital Edouard Herriot (Other)
Other Study IDs: CPP 2012-052B
Record Dates: First submitted 2013-02-09; First posted 2013-02-21 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Pain
Keywords: Analgesia Nociception Index; ANI
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to evaluate the performance of Analgesia/Nociception Index (ANI) measured at the end of surgery for the prediction of immediate postoperative pain in postoperative care unit in adult patients undergoing general anesthesia.

DETAILED DESCRIPTION:
Assessment of the performance of ANI to predict immediate postoperative pain on a 0-10 numerical rating scale (NRS) >3 by building a receiver operating characteristic curve.

ELIGIBILITY:
Inclusion Criteria:

* adult
* ear-nose-throat or orthopedic surgical procedures
* halogenated and remifentanil-based general anesthesia

Exclusion Criteria:

* age <18 yrs or >75 yrs
* arrythmia
* administration of anticholinergic drugs or neuromuscular blockade reversal in the 20 previous minutes
* psychiatric diseases
* autonomic nervous system disorders (epilepsy)
* inability to understand the verbal rating pain scale

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients underoing surgical procedures performed on general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Analgesia/Nociception Index (ANI) receiver operating characteristic (ROC) curve area under the curve (AUC) for the prediction of immediate postoperative pain | At day 0 at the end of surgery immediately before extubation for ANI and at arrival in postoperative care unit within 10 minutes after arrival
  ROC curve AUC

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Boselli, MD, PhD, Study Director — Hôpital Edourd Herriot; Bernard Allaouchiche, Md, PhD, Study Chair — Hôpital Edouard Herriot
Locations (1):
- Édouard Herriot hospital, HCL, Lyon, Rhône, France

REFERENCES:
- [Background] Boselli E, Daniela-Ionescu M, Begou G, Bouvet L, Dabouz R, Magnin C, Allaouchiche B. Prospective observational study of the non-invasive assessment of immediate postoperative pain using the analgesia/nociception index (ANI). Br J Anaesth. 2013 Sep;111(3):453-9. doi: 10.1093/bja/aet110. Epub 2013 Apr 16. PMID 23592690
- [Derived] Boselli E, Bouvet L, Begou G, Dabouz R, Davidson J, Deloste JY, Rahali N, Zadam A, Allaouchiche B. Prediction of immediate postoperative pain using the analgesia/nociception index: a prospective observational study. Br J Anaesth. 2014 Apr;112(4):715-21. doi: 10.1093/bja/aet407. Epub 2013 Dec 8. PMID 24322571